CLINICAL TRIAL: NCT03821064
Title: Single-arm, Phase II Study Evaluating the Clinical Impact of Navigation on Delays and Racial Disparities Starting Postoperative Radiation Therapy for Adults With Locally Advanced Head and Neck Cancer: The NDURE Study
Brief Title: Single-arm Phase II Study of NDURE for Patients With HNC
Acronym: NDURE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Evan Graboyes, Assistant Professor, Department of Otolaryngology- Head and Neck Surgery, Medical University of South Carolina
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00077402
Record Dates: First submitted 2019-01-24; First posted 2019-01-29 (Actual); Results first posted 2021-02-01 (Actual); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: Cancer of Head and Neck
Keywords: Cancer; Patient Navigation
MeSH Terms: conditions — Head and Neck Neoplasms; Neoplasms | interventions — Patient Navigation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient Navigation (Experimental): 45 patients (15 African American, 30 white) will interact with a patient navigator three times over three months to identify and address barriers before they cause breakdowns in care delivery, employing resources, education, and care coordination from the day of surgery until post-operative radiation treatment begins.
  Interventions: Other: Patient Navigation

INTERVENTIONS:
Other: Patient Navigation — NDURE is a theory-based, multi-level patient navigation (PN) intervention consisting of clinic-based sessions of manualized PN to reduce barriers to care, increase HNC care delivery, and improve clinical outcomes (timely, equitable PORT). NDURE will be delivered from surgical consultation to PORT initiation (~3 months). The three in-person NDURE sessions, which are expected to take 30-60 minutes each, will coincide with the presurgical consult, hospital discharge, and 1st postoperative clinic visit. During the first session, the navigator will 1) elicit barriers and facilitators to timely PORT, 2) develop the personalized barrier reduction plan (BRP), review the BRP with the patient, caregiver, and provider, and 3) implement the BRP. At the two subsequent sessions, the navigator will review and update the BRP in an iterative, dynamic fashion, identifying new barriers and systematically tracking resolution of prior barriers until the start of PORT.

SUMMARY:
This study will evaluate whether a new patient navigation intervention can decrease delays starting post-operative radiation therapy after surgery for white and African-American head and neck cancer patients.

DETAILED DESCRIPTION:
This study will evaluate the feasibility, acceptability, preliminary clinical impact, and preliminary behavioral impact of NDURE (Navigation for Disparities and Untimely Radiation thErapy), our multi-level, theory-based navigation intervention to improve timely, equitable post-operative radiation treatment (PORT) among Head and Neck Cancer (HNC) patients. We hypothesize that NDURE will be feasible, acceptable, improve the timeliness of PORT for white and African American (AA) HNC patients and decrease disparities in delay between the two groups by improving system-, interpersonal-, and individual-level health behavior constructs.

ELIGIBILITY:
In order to be eligible to participate in this study, an individual must meet all of the following criteria:

1. Age > 18 years at the time of screening
2. Histologically or pathologically confirmed invasive squamous cell carcinoma (SCC) (or histologic variant) of the oral cavity, oropharynx (p16 positive, negative, or unknown), hypopharynx, larynx, unknown primary, paranasal sinuses, or nasal cavity.
3. American Joint Committee on Cancer (AJCC) clinical stage grouping III-IV (8th edition) for patients with SCC of the oral cavity, p16-negative oropharynx, hypopharynx, larynx, paranasal sinuses, and nasal cavity; or AJCC clinical stage grouping III-IV (7th edition) for patients with p16-positive SCC of the oropharynx or unknown primary.
4. No prior exposure to radiation therapy, with or without concurrent chemotherapy, for treatment of HNSCC in the definitive or adjuvant therapy settings
5. Plan for curative intent surgery at MUSC
6. Plan for PORT (at MUSC or non-MUSC) with or without concurrent chemotherapy following curative intent surgery

An individual who meets any of the following criteria will be excluded from participation in this study:

1. Self-identified Hispanic ethnicity
2. Presence of cognitive impairment that precludes participation as determined by oncology provider
3. Prior radiation therapy for HNC
4. Failure to undergo curative intent surgery at MUSC
5. Lack of indication for PORT (with or without concurrent chemotherapy) per National Comprehensive Cancer Network (NCCN) Guidelines based on final pathologic evaluation of adverse features and AJCC pathologic stage grouping

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2019-06-03 (Actual); Primary Completion 2019-11-21 (Actual); Study Completion 2019-11-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Evan Graboyes, MD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ohlstein JF, Brody-Camp S, Friedman S, Levy JM, Buell JF, Friedlander P. Initial Experience of a Patient Navigation Model for Head and Neck Cancer. JAMA Otolaryngol Head Neck Surg. 2015 Sep;141(9):804-9. doi: 10.1001/jamaoto.2015.1467. PMID 26313895
- [Background] Cramer JD, Speedy SE, Ferris RL, Rademaker AW, Patel UA, Samant S. National evaluation of multidisciplinary quality metrics for head and neck cancer. Cancer. 2017 Nov 15;123(22):4372-4381. doi: 10.1002/cncr.30902. Epub 2017 Jul 20. PMID 28727137
- [Background] Huang J, Barbera L, Brouwers M, Browman G, Mackillop WJ. Does delay in starting treatment affect the outcomes of radiotherapy? A systematic review. J Clin Oncol. 2003 Feb 1;21(3):555-63. doi: 10.1200/JCO.2003.04.171. PMID 12560449
- [Background] Graboyes EM, Garrett-Mayer E, Ellis MA, Sharma AK, Wahlquist AE, Lentsch EJ, Nussenbaum B, Day TA. Effect of time to initiation of postoperative radiation therapy on survival in surgically managed head and neck cancer. Cancer. 2017 Dec 15;123(24):4841-4850. doi: 10.1002/cncr.30939. Epub 2017 Aug 25. PMID 28841234
- [Background] Graboyes EM, Garrett-Mayer E, Sharma AK, Lentsch EJ, Day TA. Adherence to National Comprehensive Cancer Network guidelines for time to initiation of postoperative radiation therapy for patients with head and neck cancer. Cancer. 2017 Jul 15;123(14):2651-2660. doi: 10.1002/cncr.30651. Epub 2017 Feb 27. PMID 28241092
- [Background] Divi V, Chen MM, Hara W, Shah D, Narvasa K, Segura Smith A, Kelley J, Rosenthal EL, Porter J. Reducing the Time from Surgery to Adjuvant Radiation Therapy: An Institutional Quality Improvement Project. Otolaryngol Head Neck Surg. 2018 Jul;159(1):158-165. doi: 10.1177/0194599818768254. Epub 2018 Apr 10. PMID 29631478

RESULTS

PARTICIPANT FLOW:
Groups:
- NDURE (Patient Navigation): NDURE is a theory-based, multi-level patient navigation (PN) intervention consisting of clinic-based sessions of manualized PN to reduce barriers to care, increase HNC care delivery, and improve clinical outcomes (timely, equitable PORT). NDURE will be delivered from surgical consultation to PORT initiation (~3 months). The three in-person NDURE sessions, which are expected to take 30-60 minutes each, will coincide with the presurgical consult, hospital discharge, and 1st postoperative clinic visit. During the first session, the navigator will 1) elicit barriers and facilitators to timely PORT, 2) develop the personalized barrier reduction plan (BRP), review the BRP with the patient, caregiver, and provider, and 3) implement the BRP. At the two subsequent sessions, the navigator will review and update the BRP in an iterative, dynamic fashion, identifying new barriers and systematically tracking resolution of prior barriers until the start of PORT.
Period: Overall Study
Arm/Group | NDURE (Patient Navigation)
Started | 11
Completed | 10
Not Completed | 1
Not completed — did not meet study eligibility criteria of needing adjuvant radiation per NCCN guidelines on path | 1

BASELINE CHARACTERISTICS:
Arm/Group | NDURE (Patient Navigation)
Number analyzed (Participants) | 10
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 58 [46.75 to 71.25]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 7
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Percent of Patients With a Delay Starting Post-Operative Radiation Treatment
Description: Percent of patients who start PORT >6 weeks after surgery. Initiation of postoperative PORT > 6 weeks after surgery is defined as more than 42 calendar days from the time of the definitive surgical resection to the initiation of radiation therapy. In situations in which the surgical management of the primary tumor and the neck are staged (i.e. occur on two different calendar days), the date of the surgery for the primary tumor will be used. In situations in which an additional surgical resection is required (e.g. re-resection of positive margins to clear residual disease), the date of the earlier (i.e. attempted definitive) surgical procedure will be used to determine the target start date for PORT.
Time Frame: 6 weeks
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | Patient Navigation
Number analyzed (Participants) | 10
Participants | 4

2. Secondary Outcome: Percent Difference in PORT Delay Between White and AA HNC Patients.
Description: The difference in the rate of initiation of PORT > 6 weeks after surgery between white and AA HNC patients (i.e., the difference in the percentage of white and AA participants who initiate PORT >6 weeks after surgery)
Time Frame: 6 weeks
Population: ITT
Measure: Number; unit: percentage of participants
Arm/Group | Patient Navigation
Number analyzed (Participants) | 10
percentage of participants | 9.6

3. Secondary Outcome: Median Difference in Time-to-PORT, in Days, Between White and African American HNC Patients
Description: Median difference in time-to-PORT, defined as the difference in number of days from surgery to initiation of PORT between white and AA HNC patients
Time Frame: 12 weeks
Population: ITT
Measure: Median (Standard Deviation); unit: days
Arm/Group | Patient Navigation
Number analyzed (Participants) | 10
days | 0 (17.9)

4. Secondary Outcome: Time-to-PORT
Description: Days between surgery and the start of PORT is defined as the time, in days, between the date of definitive surgical resection to the initiation of radiation therapy. All of the criteria used to adjudicate the date of the definitive surgical procedure described for the primary outcome measure will be applied to this measure.
Time Frame: 12 weeks
Population: ITT
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Patient Navigation
Number analyzed (Participants) | 10
days | 42 [36.6 to 49.6]

5. Secondary Outcome: Percent of Patients With Pre-Surgical Radiation Consultation
Description: Percent of patients with pre-surgical radiation consultation as defined as the attendance by the patient at a consultation with a radiation oncologist (at MUSC or elsewhere) prior to surgery to discuss RT in the definitive or adjuvant setting.
Time Frame: 12 weeks
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | Patient Navigation
Number analyzed (Participants) | 10
Participants | 3

6. Secondary Outcome: Percent of Patients With On-time Pre-Radiation Therapy Dental Extractions
Description: Percent of patients with on-time dental extractions, defined as the extraction of teeth prior to discharge from the index hospitalization for the definitive surgical procedure. Patients who are edentulous are not evaluable for this measure.
Time Frame: 12 weeks
Population: ITT- modified (the endpoint is only evaluable for dentate patients and 3 patients were edentulous and thus not evaluable for the endpoint)
Measure: Count of Participants; unit: Participants
Arm/Group | Patient Navigation
Number analyzed (Participants) | 7
Participants | 6

7. Secondary Outcome: Percent of Patients Surgery to Pathology Reports </= 7 Days
Description: Surgery to Pathology Report </= 7 days is defined as the production of the pathology report from the definitive surgical procedure within the electronic medical record (EMR) within 7 calendar days of the definitive surgical procedure. Addenda to the pathology report at the request of the HNC team (e.g. tumor p16 status) are not counted in this measure.
Time Frame: 12 weeks
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | Patient Navigation
Number analyzed (Participants) | 10
Participants | 8

8. Secondary Outcome: Percent of Patients With Referral to PORT Within 10 Days of Surgery
Description: Percent of patients with surgery to PORT referral </= 10 days, defined as the placement of a referral for PORT, at MUSC or elsewhere, within 10 calendar days of the definitive surgical procedure.
Time Frame: 12 weeks
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | Patient Navigation
Number analyzed (Participants) | 10
Participants | 8

9. Secondary Outcome: Percent of Patients With RT Consult Within 10 Days of RT Referral
Description: Percent of patients with RT Referral to Consult </= 10 days, defined as the evaluation of the patient at a postoperative consultation with a radiation oncologist within 10 calendar days of the referral being placed (or postoperative appointment being scheduled in cases in which care has been established and the return visit is no longer a consultation). The consultation may occur in the clinic or the hospital depending upon clinical circumstances.
Time Frame: 12 weeks
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | Patient Navigation
Number analyzed (Participants) | 10
Participants | 6

10. Secondary Outcome: Percent of Patients With Initiation of RT Within 21 Days of Consultation
Description: Percent of patients with RT Consult to Initiation </= 21 days, defined as the initiation of PORT within 21 calendar days of the patient being evaluated by a radiation oncologist for PORT.
Time Frame: 12 weeks
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | Patient Navigation
Number analyzed (Participants) | 10
Participants | 3

11. Secondary Outcome: Barriers Resolved
Description: The number of barriers identified by the navigator that are resolved during the NDURE intervention, as determined by the navigator log.
Time Frame: 12 weeks
Population: ITT
Measure: Mean (Standard Deviation); unit: barriers
Arm/Group | Patient Navigation
Number analyzed (Participants) | 10
barriers | 2.4 (1.7)

12. Secondary Outcome: Change in Self-Efficacy in Cancer Care Score From Baseline to End-of-study
Description: The Communication and Attitudinal Self-Efficacy Scale for Cancer-12 (CASE-cancer) measures self-efficacy within the context of productive communication and positive attitude for cancer patients. It is a psychometrically sound tool that may provide new information on important mediating factors of cancer care. The response scale ranges from 1 to 4 points (1= strongly disagree, 2=slightly disagree, 3=slightly agree, 4=strongly disagree). The twelve question scale is divided into 3 domains with 4 questions each. Scores from these subscales are added to compute a total score ranging from 12-48. Higher values represent a more positive attitude.
Time Frame: 12 weeks
Population: ITT- 3 participants did not complete the questionnaire
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Patient Navigation
Number analyzed (Participants) | 7
score on a scale | -1.86 (14.79)

13. Secondary Outcome: Barriers Unresolved
Description: The number of barriers identified by the navigator that are not resolved during the NDURE intervention, as determined by the navigator log.
Time Frame: 12 weeks
Population: ITT
Measure: Mean (Standard Deviation); unit: unresolved barriers
Arm/Group | Patient Navigation
Number analyzed (Participants) | 10
unresolved barriers | 0 (0)

14. Secondary Outcome: Percent of Eligible Participants Who Accrue to NDURE
Description: Percent of eligible participants who accrue to NDURE, defined as a participant who meets all inclusion criteria and no exclusion criteria
Time Frame: 13 months
Population: eligible patients
Measure: Number; unit: percentage of eligible participants
Arm/Group | Patient Navigation
Number analyzed (Participants) | 13
percentage of eligible participants | 84.6

15. Secondary Outcome: Percentage of Enrolled Participants Who Complete NDURE
Description: Percentage of enrolled participants who complete NDURE, defined as eligible patients who complete the baseline assessment, at least two NDURE intervention sessions, and the final follow-up assessment
Time Frame: 13 months
Population: ITT
Measure: Number; unit: percentage of enrolled participants
Arm/Group | Patient Navigation
Number analyzed (Participants) | 10
percentage of enrolled participants | 70

16. Secondary Outcome: Navigation Session Completion
Description: The number of NDURE navigation sessions completed by a participant
Time Frame: 12 weeks
Population: ITT
Measure: Mean (Standard Deviation); unit: NDURE sessions
Arm/Group | Patient Navigation
Number analyzed (Participants) | 10
NDURE sessions | 3 (0)

17. Secondary Outcome: Navigator Caseload
Description: The number of simultaneous cases (on-trial participants) being navigated by the NDURE navigator
Time Frame: 13 months
Population: ITT
Measure: Mean (Full Range); unit: NDURE participants
Arm/Group | Patient Navigation
Number analyzed (Participants) | 10
NDURE participants | 3 [1 to 4]

18. Secondary Outcome: Navigator Time Allocation (Direct)
Description: The time (in minutes), that the NDURE navigator spends directly interacting with the patient to identify and address barriers to timely, equitable postoperative radiation therapy
Time Frame: 12 weeks
Population: ITT
Measure: Mean (Full Range); unit: minutes
Arm/Group | Patient Navigation
Number analyzed (Participants) | 10
minutes | 100 [60 to 135]

19. Secondary Outcome: Navigator Time Allocation (Indirect)
Description: The time (in minutes), that the navigator spends generating and enacting each Barrier Reduction Plan that is not directly interacting with the patient
Time Frame: 12 weeks
Population: ITT
Measure: Mean (Full Range); unit: minutes
Arm/Group | Patient Navigation
Number analyzed (Participants) | 10
minutes | 120 [90 to 180]

20. Secondary Outcome: Satisfaction With the Interpersonal Relationship With the Navigator Scale Score
Description: The PSN-I measures the satisfaction with the interpersonal relationship with the patient navigator. The PSN-I score is defined as the total score of this 9-item scale. The total score ranges from 9 (minimum) to 45 (maximum); higher scores represent a better outcome (greater satisfaction with the interpersonal relationship with the navigator).
Time Frame: 12 weeks
Population: ITT- two participants failed to return the end of study questionnaire
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Patient Navigation
Number analyzed (Participants) | 8
units on a scale | 39.1 (8.7)

21. Secondary Outcome: Satisfaction With Logistical Aspects of Navigation Scale Score
Description: This 26-item scale measures the satisfaction of the logistical aspects of PN. The total score of the measure ranges from 0 (minimum) to 78 (maximum); higher scores represent a better outcome (greater satisfaction with the logistical aspects of navigation).
Time Frame: 12 weeks
Population: ITT- two participants failed to turn in end-of study questionnaires
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Patient Navigation
Number analyzed (Participants) | 8
units on a scale | 43.1 (25.8)

22. Secondary Outcome: Change in Care Transition Measure-15 (CTM-15) Score From Baseline to End-of-study
Description: Care Transition Measure-15 (CTM-15) is a validated, psychometrically sound 15-item, unidimensional measure of care transitions across the healthcare system that is consistent with the concept of patient-centeredness and useful from an organization perspective for the purpose of performance measurement and quality improvement. Items are rated on a 4-point Likert scale from 'Strongly Disagree' (1) to 'Strongly Agree' (4). The CTM-15 score is calculated as the mean score (the summed score from each question divided by the total number of questions) with a linear transformation to 100. Scores range from 0-100; higher scores reflect more care integration and better care transitions.
Time Frame: 12 weeks
Population: ITT- 3 did not complete the questionnaire
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Patient Navigation
Number analyzed (Participants) | 7
score on a scale | 39.5 (11.5)

23. Secondary Outcome: Change in Interpersonal Support Evaluation List-12 (ISEL-12) Score From Baseline to End-of-study
Description: The ISEL-12 is a validated, 12-item assessment of three subscales (appraisal, belonging, and tangible) that has been used to assess support in prior PN studies. Items are rated on a 4-point Likert scale from 'Definitely False' (1) to 'Definitely True' (4). The total score is calculated by summing scores across all items (with reverse coding for items 1, 2, 7, 8, 11, 12). Scores range from 12-48. Higher scores indicate more support.
Time Frame: 12 weeks
Population: ITT- 1 did not complete baseline questionnaire and 2 different participants did not complete end of study questionnaire leaving 7 evaluable paired pre-post data points
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Patient Navigation
Number analyzed (Participants) | 7
score on a scale | -0.14 (7.47)

24. Secondary Outcome: Change in Perceived Susceptibility Questionnaire Score From Baseline to End-of-study
Description: The Perceived Susceptibility Questionnaire is modified version of a validated 3-item perceived susceptibility subscale for mammography screening to assess perceived susceptibility for delays starting PORT after HNC surgery. Items are rated on a 5-point Likert scale. Scores range from 3-15 with higher scores indicating higher perceived susceptibility.
Time Frame: 12 weeks
Population: 4 participants did not complete a post questionnaire
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Patient Navigation
Number analyzed (Participants) | 6
score on a scale | -0.67 (1.03)

25. Secondary Outcome: Change in Illness Perception Questionnaire-Revised (IPQ-R) Consequences Subscale Score From Baseline to End-of-study
Description: The IPQ-R consequences subscale is easily modifiable to asses disease-specific perceived severity. The IPQ-R is a validated assessment of a patient's self-representation of the health consequences of their illness. There are 6 Items; each is rated using a 5-point Likert scale from 'Strongly Disagree' (1) to 'Strongly Agree' (5). The score is calculated by summing across all items (with reverse coding for item 3). Scores range from 5 to 30. Higher scores indicate a greater degree of perceived severity of the illness.
Time Frame: 12 weeks
Population: ITT- 3 participants did not complete the questionnaire
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Patient Navigation
Number analyzed (Participants) | 7
score on a scale | -0.17 (3.06)

26. Secondary Outcome: Change in Perceived Barriers Score From Baseline to End-of-study
Description: The Perceived Barriers Questionnaire is a self-report measure of the presence/absence of pre-specified barriers to cancer care (yes/no). The questionnaire has been used extensively to assess perceived barriers in prior PN studies. Scores range from 0-29; higher scores reflect a greater number of barriers to care
Time Frame: 12 weeks
Population: ITT- 3 did not complete post-treatment questionnaire
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Patient Navigation
Number analyzed (Participants) | 7
score on a scale | 2.2 (3.46)

ADVERSE EVENTS:
Time Frame: from baseline to initiation of postoperative radiation therapy
Description: the specific period of time is variable in this study, with end-of study defined as the initiation of postoperative radiation therapy (or 12 weeks if PORT is never started)
Arm/Group | Patient Navigation
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Informed Consent Form (2019-09-18): https://cdn.clinicaltrials.gov/large-docs/64/NCT03821064/ICF_001.pdf
  • Study Protocol and Statistical Analysis Plan (2019-07-31): https://cdn.clinicaltrials.gov/large-docs/64/NCT03821064/Prot_SAP_002.pdf